CLINICAL TRIAL: NCT01826435
Title: Improving Medication Adherence in Hypertensive Patients
Acronym: HTNmobile
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator was not clear on how best to proceed with this project.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00043793
Record Dates: First submitted 2013-04-04; First posted 2013-04-08 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic Intervention (Experimental): Over the three months, participants will receive a technology intervention. This will include text or email encounter notifications associated with appropriate mobile or online self-management information for medication adherence and behavior change.
  Interventions: Behavioral: Electronic Intervention

INTERVENTIONS:
Behavioral: Electronic Intervention — Patients will be able to receive the intervention notifications over the electronic/multimedia mode they prefer; selecting either text messaging/mobile web and/or email/online web. Text message or email alerts with an included uniform resource locator (URL) link to the specified mobile or online web site will be utilized to notify patients of a pending encounter available on mobile. Topics that will be addressed in the intervention include medication and side effects, social support, hypertension knowledge, memory and smoking. All intervention encounters that are designed to collect responses from the patient will require the patient to supply credentials before responding to the encounter; thus, ensuring privacy of the patient session, as well as patient-specific tracking of responses.

SUMMARY:
The study team is proposing a single arm intervention to test the effect of an electronic intervention on medication use among individuals with a prescription for hypertension/high blood pressure. The investigator proposes that technology like text messaging, email, web applications and mobile apps with proven, nurse intervention scripts, will lead to significant, cost-effective improvements in hypertension medication use.

DETAILED DESCRIPTION:
The intervention will incorporate a scalable electronic intervention using Email/Web Apps and Short Message Service (SMS)/Mobile Web Apps. The study team will examine the participants' responses to the electronic encounters in the technology-only intervention throughout the 3-month study timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the primary care clinic for the past 6 months
* New or existing prescription for hypertension
* Poorly controlled mean systolic blood pressure (SBP) in the last 12 months (>140/90 Hg)

Exclusion Criteria:

* Hospitalized for a stroke, myocardial infarction, coronary artery revascularization in the past 3 months,
* Diagnosis of metastatic cancer;
* Active diagnosis of psychosis or dementia documented in medical record;
* Does not have access to the appropriate technology required
* Is not willing to use said device to receive notifications for the study;
* Does not live independently (assisted living or nursing home residents) or otherwise institutionalized or receiving home health care
* Severely impaired hearing, vision or speech (unless technological aides allow them full functionality)
* Planning to leave the area or change primary care clinics prior to the anticipated end of participation;
* Unable to read and understand spoken English
* Participation in another cardiovascular disease (CVD) study
* Another household member enrolled in study;
* Arm size > 50cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of Days Covered (PDC) | 3 months
  Proportion of Days Covered (PDC), a Pharmacy Quality Alliance (PQA)-recommended metric for estimation of medication adherence for patients using chronic medications, will be used to identify the percentage of patients taking medications in a particular drug class with high adherence (PDC > 80% for the individual). Participants with a PDC ≤0.8 will be categorized as having "poor" adherence, and those with a PDC >0.8 will be categorized as having "good" adherence. For analyses, the PDC will be dichotomized at 0.8 (PDC >0.8) over the entire 3 month follow-up, yielding a single assessment of pill refill adherence that will be used as the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System Clinic, Durham, North Carolina, United States